CLINICAL TRIAL: NCT01533298
Title: A Randomized, Open, Multicenter, Compared Phase III Trial to Evaluate the Safety, Efficacy of CombiflexOmega Peri and SmofKabiven Peripheral in Postoperative Patients Requiring Parenteral Nutrition
Brief Title: A Safety, Efficacy Study of CombiflexOmega Peri Versus SmofKabiven Peripheral in Patients With Parenteral Nutrition
Acronym: OMEGA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Life Science (Industry)
Responsible Party: Sponsor
Organization: JW Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CW-CFO-301
Record Dates: First submitted 2012-01-18; First posted 2012-02-15 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Parent

ARMS (2):
- CombiflexOmega peri (Experimental)
  Interventions: Drug: CombiflexOmega peri
- SmofKabiven peripheral (Active Comparator)
  Interventions: Drug: SmofKabiven peripheral

INTERVENTIONS:
Drug: CombiflexOmega peri — intravenously over 3 days infusion
  Arms: CombiflexOmega peri
Drug: SmofKabiven peripheral — intravenously over 3 days infusion
  Arms: SmofKabiven peripheral

SUMMARY:
The purpose of this study is to compare the safety and efficacy of CombiflexOmega peri in comparison to SmofKabiven peripheral in postoperative patients requiring parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 and older
* Patients are expected to require PN for more than 3 days
* Patients who voluntarily signed the consent form

Exclusion Criteria:

* Patients are expected difficult to survive more than 3 days
* Pregnant or breast-feeding women
* BMI > 30 kg/m2
* Patients with severe blood coagulation disorders
* Patients with congenital amino acid metabolism disorders
* Patients with acute shock
* Patients with uncontrollable diabetes mellitus
* Patients with hemophage syndrome
* Patients with hypopotassemia (K < 3.0mEq/L)
* Patients having the history of myocardial infarction
* Patients reported the following laboratory value

  * fasting TG > 250mg/dl, TC > 300mg/dl
  * ALT/AST ≥ 2×ULN, Bilirubin ≥ 3mg/dl (Exception : patients with periampullary carcinoma including biliary tract or pancreas)
  * Creatinine ≥1.5mg/dl
  * Ca > 11.2mg/dl, Na ≥ 145mEq/L, Mg ≥ 2.1mEq/L, K ≥ 5.5mEq/L
* Patients having hypersensitivity to any peanut-, fish-, soy-, egg protein, or investigational drug
* Patients having the history of drug or alcohol abuse
* General contraindications to infusion therapy: acute pulmonary oedema, hyperhydration, cardiac decompensation
* Patients are in unstable conditions
* Patients with difficult peripheral intravenous
* Patients with parenteral nutrition within 7 days prior to start of the trial
* Participation in another clinical study with an investigational drug or an investigational medical device within 28 days prior to start of study
* Patients judged to be unsuitable for this trial by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Comparison of adverse drug reaction | 4days

SECONDARY OUTCOMES:
Changes of laboratory parameters (biochemistry, hematology, coagulation) | 5days
Changes of vital signs | 5days

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea